CLINICAL TRIAL: NCT02194192
Title: Prophylaxis Ephedrine or Ondansetron Prevents Hypotension After Spinal Anesthesia for Cesarean Section; a Randomized, Double Blinded, Placebo Controlled Trial
Brief Title: Prophylaxis Ephedrine or Ondansetron Prevents Hypotension After Spinal Anesthesia for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 810/2556(EC2); (IO)R015731034 (Other Grant/Funding Number: Faculty of medicine Siriraj Hospital, Mahidol University)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural
Keywords: prevention of hypotension; spinal anesthesia; cesarean section; ephedrine; ondansetron
MeSH Terms: interventions — Ondansetron; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group E (Experimental): Ephedrine 10 mg in Normal Saline 10 ml
  Interventions: Drug: Ephedrine
- Group O (Active Comparator): Ondansetron 8 mg in Normal saline 10 ml
  Interventions: Drug: Ondansetron
- Group P (Placebo Comparator): Normal saline 10 ml
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Normal saline 10 ml
  Arms: Group P
Drug: Ondansetron — Ondasetron 8 mg IV after spinal anesthesia
  Arms: Group O
Drug: Ephedrine — Ephedrine 10 mg IV after spinal anesthesia
  Arms: Group E

SUMMARY:
Maternal hypotension after spinal anesthesia in parturients undergoing cesarean section is a very common problem leading to several complications to both patients and their babies. It can cause maternal discomfort, lightheadedness, nausea and vomiting. The most important complication is the decreasing blood flow to babies; which may lead to fetal acidosis.

Many interventions has been studied in order to prevent hypotension after spinal anesthesia in cesarean section e.g., fluid loading: colloid vs crystalloid, medications: ephedrine, phenylephrine, and metaraminol, etc. The recent study showed ondansetron (the antiemetic drug) can be effectively used to prevent hypotension after spinal anesthesia in normal patients or parturients. The action of ondansetron is believed to inhibit Bezold-Jarish reflex.

This aim of this study is to compare the efficacy of ephedrine and ondansetron in the prevention of maternal hypotension after spinal anesthesia in cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Elective cesarean section
* Patient accept spinal anesthesia
* ASA classification I-II
* Term, Singleton pregnancy
* Understand all process in this study

Exclusion Criteria:

* DM any type that not the gestational DM
* Hypertensive disorder
* BMI>40
* Complicated pregnancy such as placenta previa, preeclampsia
* Allergic to study drugs
* Long QT syndrome
* Contraindication to spinal anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Comparing efficacy of ondansetron to ephedrine in the prevention of hypotension. | After spinal block to until baby delivered
  Ondansetron or ephedrine will be given immediately after spinal anesthesia, then record blood pressure and heart rate one-minutely until delivery.

SECONDARY OUTCOMES:
Maternal symptom: Nausea and vomiting after spinal anesthesia | After spinal anesthesia until baby delivered

OTHER OUTCOMES:
Apgar score | one minute and five minute after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Sahoo T, SenDasgupta C, Goswami A, Hazra A. Reduction in spinal-induced hypotension with ondansetron in parturients undergoing caesarean section: a double-blind randomised, placebo-controlled study. Int J Obstet Anesth. 2012 Jan;21(1):24-8. doi: 10.1016/j.ijoa.2011.08.002. Epub 2011 Nov 18. PMID 22100822
- [Background] Owczuk R, Wenski W, Polak-Krzeminska A, Twardowski P, Arszulowicz R, Dylczyk-Sommer A, Wujtewicz MA, Sawicka W, Morzuch E, Smietanski M, Wujtewicz M. Ondansetron given intravenously attenuates arterial blood pressure drop due to spinal anesthesia: a double-blind, placebo-controlled study. Reg Anesth Pain Med. 2008 Jul-Aug;33(4):332-9. doi: 10.1016/j.rapm.2008.01.010. PMID 18675744
- [Background] Lee A, Ngan Kee WD, Gin T. Prophylactic ephedrine prevents hypotension during spinal anesthesia for Cesarean delivery but does not improve neonatal outcome: a quantitative systematic review. Can J Anaesth. 2002 Jun-Jul;49(6):588-99. doi: 10.1007/BF03017387. PMID 12067872
- [Background] Cyna AM, Andrew M, Emmett RS, Middleton P, Simmons SW. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD002251. doi: 10.1002/14651858.CD002251.pub2. PMID 17054153
- [Background] Lee A, Ngan Kee WD, Gin T. A dose-response meta-analysis of prophylactic intravenous ephedrine for the prevention of hypotension during spinal anesthesia for elective cesarean delivery. Anesth Analg. 2004 Feb;98(2):483-490. doi: 10.1213/01.ANE.0000096183.49619.FC. PMID 14742392